CLINICAL TRIAL: NCT06209502
Title: Q-Index: A Proof of Concept Investigation Towards Monitoring the Health-related Quality of Life of Parkinson's Disease Patients Using Wearable and Portable Devices.
Brief Title: Quality-of-Life Index (Q-Index)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Koios Care (Industry)
Responsible Party: Sponsor
Other Study IDs: KC-QI-2023
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: Smartwatch; Smartphone; Quality of life; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Population A: Parkinson's disease patients between H&Y stages 1.5 and 3
- Population B: Early Parkinson's disease patients of H&Y stage 1
- Population C: Healthy controls

SUMMARY:
The main objective of this observational study is to use commonly-used connected objects (smartphones and smartwatches) to remotely assess and monitor the health-related quality of life (HrQoL) of people with Parkinson's disease at different stages of progression.

DETAILED DESCRIPTION:
The main objective of this observational study is to use commonly-used connected objects (smartphones and smartwatches) to remotely assess and monitor the health-related quality of life (HrQoL) of people with Parkinson's disease at different stages of progression.

The study takes place in hospitals in Belgium. The study populations are as follows: up to 100 patients between stages H&Y 1.5 and 3 (population A), up to 15 patients with early-stage Parkinson's disease H&Y 1 (population B), and up to 15 healthy controls (population C). The duration of the study is approximately 9 months, between September 2023 and November 2024, and will include a baseline clinical assessment (month 0), the first follow-up (month 4) and the second follow-up (month 8).

The main objective is to build an algorithm capable of remotely assessing the health-related quality of life (HrQoL) of patients belonging to population A. This objective will be achieved by formulating and estimating the quality of life index (Q-index) based on continuously and passively recorded data from commercially available wearable devices (an Android smartwatch and a smartphone). The secondary objective is to determine whether the Q index is sufficiently sensitive to monitor the quality of life of people who are in the early stages of the disease (population B). A group of healthy control subjects (population C) will be used to identify the range of Q index values corresponding to healthy and PD populations.

To achieve this objective, we will compare the information extracted from connected devices (micro-indicators) with the responses of participants to questionnaires and clinical tests aimed at evaluating PROMs (patient-related outcome measures). The list of data collected is included in the following table.

To calculate the Q index, we plan to use a combination of several micro-indicators, each acting as a surrogate for the subject's ability to effectively perform certain activities of daily living; communication, sleep, eating, sociability and physical independence. An example of a micro-indicator is Plate-to-Mouth1 (PtM), which measures the individual's eating behavior by estimating the time required to transfer a quantity of food ready to be consumed, from the plate to the mouth.

The ability to accurately monitor health-related quality of life (HrQoL) characteristics will be assessed initially by examining how each micro-indicator correlates with appropriate items from validated questionnaires such as the Health-Related Quality of Life Questionnaire. Parkinson's disease, called PDQ-39. For example, eating behavior (and more specifically Plate-to-Mouth) is associated with upper limb sluggishness and is linked to items 11, 12, 13, 14 and 16 of the PDQ-39. After assessing each micro-indicator, the combined ability of the Q index to monitor HrQoL as a whole will be realized by comparing it to scores and subscores from validated PROMs scales, such as the PDQ-39.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 30 and 75
* Agree to download and install the Koios Care application to their personal Android smartphone.
* People diagnosed with idiopathic PD based on the MDS-PD criteria. The diagnosis must be confirmed by bradykinesia plus one of the other cardinal signs (resting tremor, rigidity or postural instability not caused by primary visual, vestibular, cerebellar, or proprioceptive dysfunction) being present, without any other known or suspected cause of Parkinson's Disease.

  o PD patients that are under the effects of a Deep Brain Stimulation (DBS) device or a levodopa pump (duodopa or lecigimon). Given that all other conditions are also met.
* Score between one-and-a-half (1.5) and three (3) at the H&Y rating scale in the "ON" state (population A)
* Score of one (1) at the H&Y rating scale in the "ON" state (population B)

Exclusion Criteria:

* The candidate cannot speak or comprehend the French/Dutch (depending on the clinical site s/he belongs to) language at a sufficient level.
* The reluctance of the candidate or her/his inability to provide written consent (e.g., due to mental health problems or severe physical disabilities).
* The candidate is not an Android smartphone owner and user for at least six (6) months.
* The candidate's Android smartphone is not compatible with the Koios Care application.
* The candidate suffers from dementia as judged by the investigator. For this we will use MMSE score with a cut-off value ≥ 24.
* The candidate has exhibited uncontrolled/extreme measures of depression as judged by the expert investigator, e.g., self-harm, suicide attempts or patient admitted to the hospital for a similar reason.

  -- If the participant develops such behavior or s/he is admitted to the hospital for the above reasons during the study, then the candidate is immediately removed from the study.
* Any Parkinson's disease-related feature or symptom that could interfere with the study conduct and results as assessed by the investigator.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruitment process for Parkinson's Disease patients begins during a consultation taking place in one of the three participating clinics. Specifically, a member of the medical team informs the patient about the ongoing study, including but not limited to, its goals, the technology, and the timeline of the study.
  The recruitment of a Parkinson's Disease patient also appears as an opportunity to recruit healthy participants. Specifically, the study targets members of the close circle of the patient, i.e., age-matched friends and close family members. It should be noted that to avoid recruitment bias (e.g., the partner of the patient stays home to support their patient partner), the partner of the patient is left as the emergency (low recruitment rate for healthy controls) recruitment scenario. In addition, the recruitment procedure for healthy controls will be supported by wall posters in the hospital campus and web advertising.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary objective | Clinical assessments are collected in the clinic at month 0, month 4 and month 8 of the study. Moreover, two self-assessment questionnaires are collected remotely (a) once per month, and (b) once per week.
  Primarily, this longitudinal study targets patients with Parkinson's Disease between the stages of one-and-a-half (1.5) and three (3) in the Hoehn & Yahr scale (in the context of this study; population A). By considering the aforementioned population, the primary objective is to build an algorithm towards the remote assessment of the individuals' Health-related QoL (HrQoL). This is to be achieved by formulating and estimating the Quality-of-Life index (Q-index) based on continuously and passively recorded data from commercially available wearable and portable technology (i.e., an Android smartwatch and an Android smartphone).

SECONDARY OUTCOMES:
Secondary objective | Clinical assessments are collected in the clinic at month 0, month 4 and month 8 of the study. Moreover, two self-assessment questionnaires are collected remotely (a) once per month, and (b) once per week.
  Investigate whether the Q-index is sensitive enough to monitor the HrQoL of early PD patients that belong in H&Y stage 1 (population B).

OTHER OUTCOMES:
Exploratory objective 1 | Clinical assessments are collected in the clinic at month 0, month 4 and month 8 of the study. Moreover, two self-assessment questionnaires are collected remotely (a) once per month, and (b) once per week.
  Build an algorithm with the ability to predict the score of the clinical assessments regarding the progression of the disease, based on past assessments, sensor data and PROMs - populations A and B.
Exploratory objective 2 | Clinical assessments are collected in the clinic at month 0, month 4 and month 8 of the study. Moreover, two self-assessment questionnaires are collected remotely (a) once per month, and (b) once per week.
  Assess if individual fluctuations in PROMs are more accurately captured by the Q-index rather than the traditional clinical instruments of disease severity - populations A and B. A toy example can be found in Figure 1. A group of Healthy Controls (HCs), population C, will be used for further evaluation and to identify the range of values of the Q-index that correspond to the healthy and Parkinsonian populations.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Delta, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: No